CLINICAL TRIAL: NCT02289859
Title: Undermining During Cutaneous Wound Closure: a Randomized Split Wound Comparative Effectiveness Trial
Brief Title: Undermining During Cutaneous Wound Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 613430
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Wound Closure Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wound Closure with Undermining (Active Comparator): The side assigned to undermining will have undermining performed prior to wound closure in the subcutaneous plane. The amount of undermining will range from 1 cm for wounds with low tension to 2 cm for those with moderate tension. Since wound diameter will be 3 cm or less and exclude the scalp, high tension wounds are not anticipated.
  Interventions: Procedure: Wound Closure with Undermining; Procedure: Wound Closure without Undermining
- Wound Closure without Undermining (Active Comparator): One side of the wound will remain un-undermined.
  Interventions: Procedure: Wound Closure with Undermining; Procedure: Wound Closure without Undermining

INTERVENTIONS:
Procedure: Wound Closure with Undermining — The side assigned to undermining will have undermining performed prior to wound closure in the subcutaneous plane. The amount of undermining will range from 1 cm for wounds with low tension to 2 cm for those with moderate tension. Since wound diameter will be 3 cm or less and exclude the scalp, high tension wounds are not anticipated.
Procedure: Wound Closure without Undermining — One side of the wound will remain un-undermined.

SUMMARY:
The purpose of this study is to determine whether undermining during cutaneous surgery improves scar cosmesis compared to wound closure without undermining.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether undermining during cutaneous surgery improves scar cosmesis compared to wound closure without undermining. Our aims are to compare outcomes using a split wound model, where half the wound is undermined and the other half is not. This will be measured via the physician observer scar assessment scale, a validated scar instrument and via wound width. Our hypothesis is that wound undermining will result in cosmetically superior wound outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure with predicted linear closure
* Willing to return for follow up visits

Exclusion Criteria:

* Mentally handicapped
* Incarceration
* Pregnant Women
* Wounds with predicted closure length less than 3 cm
* Wounds with diameter > 3 cm
* Wounds unable to be fully closed without undermining

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Assessment of Scar on the Patient and Observer Scar Assessment Scale | 3 months
  After surgical procedure, half of the subject's wound will be closed after undermining, while the other half is closed without undermining. After 3 months, subjects will return to clinic for evaluation of the cosmesis of both types of closure techniques.

SECONDARY OUTCOMES:
Measurement of Scar Width | 3 months
  The width of the scar will be measured 1 centimeter from the midline on both sides. There is no defined width that is considered satisfactory or not satisfactory. The measurements will be compared between subjects.
Assessment of Complications | 3 months
  Noting the presence or absence of bleeding, dehiscence, infection or spitting sutures.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, M.D., Principal Investigator — University of California, Davis

REFERENCES:
- [Derived] Joo J, Pourang A, Tchanque-Fossuo CN, Armstrong AW, Tartar DM, King TH, Sivamani RK, Eisen DB. Undermining during cutaneous wound closure for wounds less than 3 cm in diameter: a randomized split wound comparative effectiveness trial. Arch Dermatol Res. 2022 Sep;314(7):697-703. doi: 10.1007/s00403-021-02280-5. Epub 2021 Sep 21. PMID 34546436
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical